CLINICAL TRIAL: NCT02685215
Title: Prognostic Factors, Morbidity, Mortality and Long Term Survival in Patients With Neuromuscular Disorders Admitted in Intensive Care Unit
Brief Title: Prognostic Factors , Morbidity and Mortality in Patients With Neuromuscular Disorders Admitted in ICU
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Centre d'Investigation Clinique et Technologique 805 (Other)
Responsible Party: Principal Investigator, Abdallah FAYSSOIL, MD PhD, Centre d'Investigation Clinique et Technologique 805
Other Study IDs: 1912677
Record Dates: First submitted 2016-01-14; First posted 2016-02-18 (Estimated); Last update posted 2019-05-16 (Actual); Status verified 2019-05

CONDITIONS: Muscular Dystrophies; Intensive Care (ICU) Myopathy
Keywords: intensive care unit; muscular dystrophy; mortality; prognosis; tracheostomy
MeSH Terms: conditions — Muscular Dystrophies; Muscular Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Muscular dystrophies are neuromuscular disorders with disability. Restrictive pulmonary failure and cardiomyopathy affect prognosis.The investigators aim to establish predictive factors for mortality and morbidity in Intensive care unit (ICU ) and to describe the long term follow up after ICU discharge.

DETAILED DESCRIPTION:
Muscular dystrophies are neuromuscular disorders with disability. Restrictive pulmonary failure and cardiomyopathy affect prognosis. Little is known about morbidity and mortality of patients with muscular dystrophies admitted in intensive care unit (ICU).The investigators aim to describe the spectrum of patients with muscular dystrophies admitted in ICU , to establish predictive factors for ICU mortality and morbidity and to describe the long term follow up after ICU discharge.

ELIGIBILITY:
Inclusion Criteria:

* admitted in ICU
* Duchenne muscular dystrophy
* Becker muscular dystrophy
* LGMD
* Steinert disease
* Pompe disease
* FSHD
* metabolic disease
* mitochondrial disease
* congenital myopathy
* others neuro-muscular diseases

Exclusion Criteria:

* brain injury
* minor patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with neuro-muscular disorders admitted in ICU since 2005
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2016-03; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
ICU mortality | 1 month

SECONDARY OUTCOMES:
tracheostomy in ICU | 1 month
predictive factors for re admission in ICU | 1 year
long term survival after ICU stay | 5 years
decline of vital capacity after ICU stay | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: abdallah Fayssoil, MDPhD, Principal Investigator — Raymond Poincare Hospital
Locations (1):
- Hopital Raymond Poincare, Garches, France

IPD SHARING:
Plan to Share IPD: No